CLINICAL TRIAL: NCT04774172
Title: Mortality and Morbidity Outcomes After Aortovascular Surgery in Patients With Marfan Syndrome: A UK Experience
Brief Title: Mortality and Morbidity Outcomes in Marfans
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Aortic Dissection Awareness UK & Ireland. (Other)
Responsible Party: Sponsor
Other Study IDs: 294022
Record Dates: First submitted 2021-02-18; First posted 2021-03-01 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Marfan Syndrome; Marfan Syndrome Cardiovascular Manifestations
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Marfan Syndrome (MFS) is a genetic disease affecting the eyes, skeleton, heart and arteries. Despite MFS affecting multiple organ systems, cardiovascular manifestations are the most serious and life threatening. Approximately 80% of adult MFS patients will have a dilated aortic root by age 40 years with aortic aneurysm and dissection the leading causes of morbidity and mortality. Improvement in diagnostics and medical and surgical interventions have increased life expectancy. However, the natural history and the influence of medical or surgical interventions in the UK population are not fully described. Further, the incidence of aortovascular surgery in this patient group is unknown as MFS is not routinely documented in the National Institute of Cardiovascular Outcome Research (NICOR) national cardiac surgery dataset and therefore, there is currently no mechanism for exploring the aortovascular outcomes for this patient group.

The investigators aim to undertake a 10-year secondary analysis of linked national data (National Institute of Cardiovascular Outcome Research (NICOR), Office of National Statistics (ONS), Hospital Episode Statistics (HES)) to identify the UK incidence and outcome of aorto-vascular surgery in patients with Marfan syndrome (MFS). This includes associated hospital length of stay, mortality and morbidity rates.

Understanding mortality alongside morbidity will allow the investigators to study further the burdens that the aortovascular manifestations may place on MFS population as well as to continuously evaluate the efficacy of either the health care system or an implemented intervention in place. Further, these metrics will be useful for the stakeholders to effectively prioritise which complications to tackle and to allocate resources toward as well as proactively manage the potential onset of a health event

DETAILED DESCRIPTION:
Marfan Syndrome (MFS) is a genetic disease affecting the eyes, skeleton, heart and arteries. Despite MFS affecting multiple organ systems, cardiovascular manifestations are the most serious and life threatening. Approximately 80% of adult MFS patients will have a dilated aortic root by age 40 years with aortic aneurysm and dissection the leading causes of morbidity and mortality. Improvement in diagnostics and medical and surgical interventions have increased life expectancy. However, the natural history and the influence of medical or surgical interventions in the UK population are not fully described. Further, the incidence of aortovascular surgery in this patient group is unknown as MFS is not routinely documented in the National Institute of Cardiovascular Outcome Research (NICOR) national cardiac surgery dataset and therefore, there is currently no mechanism for exploring the aortovascular outcomes for this patient group.

The investigators aim to undertake a 10-year secondary analysis of linked national data (National Institute of Cardiovascular Outcome Research (NICOR), Office of National Statistics (ONS), Hospital Episode Statistics (HES)) to identify the UK incidence and outcome of aorto-vascular surgery in patients with Marfan syndrome (MFS). This includes associated hospital length of stay, mortality and morbidity rates.

Understanding mortality alongside morbidity will allow the investigators to study further the burdens that the aortovascular manifestations may place on MFS population as well as to continuously evaluate the efficacy of either the health care system or an implemented intervention in place. Further, these metrics will be useful for the stakeholders to effectively prioritise which complications to tackle and to allocate resources toward as well as proactively manage the potential onset of a health event.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years old at the time of surgery
* Identified MFS in the HES database using the ICD diagnosis code Q874 between January 2010- December 2019
* Had an aorto-vascular surgery in England and Wales, as identified in the NICOR Adult Cardiac Surgery database

Exclusion Criteria:

* < 18 years old at the time of surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all eligible patients who are identified as MFS using the ICD-10 code Q874 through the National Health Service Digital (NHSD) from January 2010 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 6700 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality mortality rate 1-year after surgery. Mortality rate 1 year after aorto-vascular surgery | 1 year after surgery
  mortality rate 1-year after surgery

SECONDARY OUTCOMES:
Morbidity outcomes | within 1 year after surgery
  (i) Underlying cause of death and multiple causes of death
Morbidity outcomes | within 1 year after surgery
  Date of each Finished Consultant Episode
Morbidity outcomes | within 1 year after surgery
  Primary and secondary diagnostic codes
Morbidity outcomes | within 1 year after surgery
  Primary procedural codes
Morbidity outcomes | within 1 year after surgery
  Hospital episode length

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomews Hospital, London, United Kingdom